CLINICAL TRIAL: NCT05257876
Title: An Evidence-based Breathing Exercise Intervention Protocol for Chronic Pain Management in Breast Cancer Survivors: A Preliminary Randomized Controlled Trial
Brief Title: Breathing Exercise for Chronic Pain Management in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Darwin University (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H21089
Record Dates: First submitted 2022-02-03; First posted 2022-02-25 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain; Breast Neoplasms; Cancer Survivors
Keywords: Pain Management; Chronic Pain; Breast Neoplasms; Cancer survivors; Breathing Exercises
MeSH Terms: conditions — Chronic Pain; Breast Neoplasms; Agnosia | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Open-labelled parallel pilot RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive breathing exercise training, pain information booklet, and usual care.
  Interventions: Other: Breathing exercise
- Control group (No Intervention): Participants in the control group will receive pain information booklet and usual care.

INTERVENTIONS:
Other: Breathing exercise — Participants will receive breathing exercise training, and a 4-week self exercise
  Arms: Intervention group

SUMMARY:
The study will follow the MRC Framework to develop an evidence-based BE intervention protocol to help breast cancer survivors with better management of cancer-related chronic pain.

DETAILED DESCRIPTION:
Cancer-related chronic pain remains as a big challenge for cancer survivors, which significantly affects the quality of life of cancer survivors. Evidence suggests that pain is well managed through combination of pharmacological and non-pharmacological interventions. Among all non-pharmacological interventions, breathing exercise (BE) might have potential effect for chronic pain management in cancer survivors, but the evidence is sparse in current literature. Therefore, this study will follow the Medical Research Council Framework for Developing and Evaluating Complex intervention (the MRC Framework) to develop an evidence-based BE protocol to help with cancer-related chronic pain management in breast cancer survivors. The first two phases of the MRC Framework will be included in this study. In the first phase, an evidence-based method will be utilized to develop the BE intervention protocol. In the second phase, a pilot randomised controlled trial (RCT) will be conducted to examine the feasibility of study and the acceptability of the BE intervention by the participants as well as to preliminarily assess the effect of the BE on chronic pain management in breast cancer survivors. Semi-structured interviews will be conducted after the RCT to explore participants' experiences of participating in the study and practicing the BE.

ELIGIBILITY:
Inclusion Criteria:

1. female breast cancer survivors ≥18 years age;
2. has a confirmed diagnosis of breast cancer at stage I, II or IIIa;
3. has been experiencing pain since cancer diagnosis constantly or intermittently for ≥3 months, with the average pain intensity in the last seven days on a numerical scale ≥4/10 ("0" indicates no pain and "10" indicates the worst pain);
4. has completed active anticancer treatment (such as chemotherapy, radiotherapy, surgery) for at least three months;
5. agrees to participate in the research and is willing to give informed consent;
6. can read and understand Mandarin Chinese.

Exclusion Criteria:

1. extremely weak and unable to perform the breathing exercises;
2. mentally incapable (i.e., unable to follow the study instructions);
3. has scheduled pain management interventions, such as having a procedure or operation;
4. receiving other pain relief treatments, such as acupuncture, yoga, qigong, exercise program, etc.;
5. has any pre-existing chronic pain conditions before cancer diagnosis, such as arthritis, rheumatoid arthritis, chronic low back pain, migraines, trigeminal neuralgia, fibromyalgia, joint dysfunction, Complex Regional Pain Syndrome, endometriosis, etc.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender eligibility is based on the physical appearance.
Enrollment: 72 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
Feasibility: Time taken to recruit planned sample | Immediately after the allocation of the last subject
  The time that was taken to recruit the planned sample size of participants
Feasibility: Referral rate | Immediately after the referral of the last subject
  The number of referrals made by clinicians in different departments divided by all referrals
Feasibility: Recruitment rate | Immediately after the recruitment of the last subject
  Proportion of subjects who participated in the study from all subjects eligible for participation
Feasibility: Retention rate | At the follow-up assessment 4 weeks after the intervention completion (T3)
  Proportion of participants who completed the whole study divided by all subjects who enrolled in the study
Feasibility: Dropout rate | At the follow-up assessment 4 weeks after the intervention completion (T3)
  The number of subjects who dropped out after randomization divided by all subjects who enrolled in the study
Reasons for dropping out | Immediately once a dropout occurs
  Feedback from the dropout subjects to identify their reasons for dropping out
Feasibility of the questionnaires | At baseline (T1), immediately after the completion of the 4-week intervention (T2), and the follow-up assessment at 4 weeks after the intervention completion (T3)
  The percentage of missing values for each item of the scales used, including the Brief Pain Inventory (BPI), Quality of life Cancer Survivors Version (QOL-CSV), Functional Assessment Cancer Therapy-Breast (FACT-B), and Hospital Anxiety and Depression Scale (HADS)
Feasibility: Adherence rates | Immediately after completion of the 4-week intervention (T2)
  the percentage of BE sessions performed by participants divided by the total number of BE sessions required
Participants' feedback | Immediately after completion of the 4-week intervention (T2)
  Participants' feedback on and satisfaction with the intervention using a specifically designed feedback form
Adverse events associated with the intervention | Immediately once an adverse event occurs
  Data will be collected from the participants' BE logbooks and supplemented by information collected during weekly telephone contact

SECONDARY OUTCOMES:
Chronic pain | At baseline (T1), immediately after the completion of the 4-week intervention (T2), and the follow-up assessment at 4 weeks after the intervention completion (T3)
  Chronic pain will be measured by using the Brief Pain Inventory which measures pain intensity and pain interference with the life. For pain severity, four items are used to measure the "worst", "least", "average" and "now" with a rating scale from 0 to 10, higher number indicating the higher score in each item. For pain interference, pain is measured from 7 aspects of general activity, mood, walking, work, relations with others, sleep and enjoyment of life with a scale of 0-10, and higher score indicates severe impact of pain.
Quality of life of breast cancer survivors ( using tool 1) | At baseline (T1), immediately after the completion of the 4-week intervention (T2), and the follow-up assessment at 4 weeks after the intervention completion (T3)
  Quality of life will be measured by using the Quality of Life Cancer Survivors Version. This questionnaire contains 41 items measuring quality of life of cancer survivors from four aspects including physical well-being, psychological well-being, social well-being and spiritual well-being. The score of each item is based on a scale of 0 ( worse outcome) to 10 ( best outcome). Higher score indicates better quality of life.
Quality of Life of breast cancer survivors ( using tool 2) | At baseline (T1), immediately after the completion of the 4-week intervention (T2), and the follow-up assessment at 4 weeks after the intervention completion (T3)
  Quality of life will also be measured by using the Functional Assessment of Cancer Therapy-Breast. This questionnaire has 37 items with a 5-point Likert scale ranging from 0 to 4, a higher score indicating better QoL.
Anxiety and Depression | At baseline (T1), immediately after the completion of the 4-week intervention (T2), and the follow-up assessment at 4 weeks after the intervention completion (T3)
  Anxiety and depression will be measured by using the Hospital Anxiety and Depression Scale (HADS). This scale contains 14 items consisting of two subscales: the anxiety subscale and depression subscale with 7 items in each. The scale uses a 4-point Likert scale ranging from 0 to 3, and higher score indicates severe anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Jing-Yu (Benjamin) Tan, PhD, Principal Investigator — Charles Darwin University
Locations (1):
- The Affiliated Hospital Of Southwest Medical University, Luzhou, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
It needs to get the participants' consent if the data is shared with other researchers.

REFERENCES:
- [Derived] Wang H, Tan JB, Wang T, Liu XL, Bressington D, Zheng SL, Huang HQ. Feasibility and potential effects of breathing exercise for chronic pain management in breast cancer survivors: study protocol of a phase II randomised controlled trial. BMJ Open. 2022 Dec 14;12(12):e064358. doi: 10.1136/bmjopen-2022-064358. PMID 36517097

DOCUMENTS (1):
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT05257876/ICF_000.pdf